CLINICAL TRIAL: NCT03179553
Title: Improving Early Decisions in Neonatal Encephalopathy by Monitoring Heartbeat Variability
Brief Title: Heart Beat Variability in Neonatal Encephalopathy
Acronym: HeartBeat
Status: Active, not recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 17HH3917
Record Dates: First submitted 2017-06-06; First posted 2017-06-07 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Neonatal Encephalopathy; Asphyxia Neonatorum; Hypoxic-Ischemic Encephalopathy
MeSH Terms: conditions — Asphyxia Neonatorum; Hypoxia-Ischemia, Brain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — salivary swabs for cortisol measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HIE: Babies admitted to the neonatal unit with suspected mild, moderate or severe hypoxic ischaemic encephalopathy .
- Healthy: Babies who are inpatients in the postnatal ward, born following uncomplicated pregnancy and delivery.

SUMMARY:
This study will find out if analysing heartbeat in babies with brain injury, based on standard clinical monitors, can inform treatment decisions and monitor stress levels in real time

DETAILED DESCRIPTION:
BACKGROUND

Hypoxic ischaemic encephalopathy (HIE) is the single most common cause of death and lifelong neurodisability in term babies. Although cooling treatment improves outcomes for these babies, early identification (within six hours of birth) of 'at risk infants' remains challenging. Consequently, not all babies who need treatment will receive it and other babies receive treatment unnecessarily. Furthermore, neuroprotection from cooling may be lost if baby remains stressed during treatment, but accurate methods of measuring stress in babies are lacking.

AIMS

Primary aim:

To examine the accuracy of heartbeat variability (HRV), within six hours of birth, to predict adverse neurodevelopmental outcome at 18 to 22 months in encephalopathic babies.

Secondary aims:

* To examine the relation between heartbeat variability and stress in encephalopathic babies.
* To identify clinical interventions associated with reduced heartbeat variability in encephalopathic babies.
* To describe the trajectory of normal heartbeat variability changes in healthy term babies during the first 24 hours after birth.

METHODS

A total 140 term babies with hypoxic ischaemic encephalopathy will be recruited. The investigators will collect continuous electrocardiography (ECG) data, hourly Neonatal Pain Agitation and Sedation Scale (NPASS) and 12 hourly salivary cortisol, for the first five days after birth. Various clinical interventions, and noise and light levels that the baby is exposed to, for the first 5 days after birth will be be recorded.

The investigators will analyse the raw ECG using Matlab® with in-house algorithms to quantify specific linear and non-linear measures of HRV. All recruited encephalopathic babies will have brain magnetic resonance (MR) imaging and spectroscopy using harmonised protocols and neurodevelopmental assessment, as a part of clinical care, or as a part of MR biomarker studies. This data will be collected and used for the Heartbeat study to examine the association between heart rate variability with brain injury and neurodevelopmental outcome.

In addition, the investigators will collect the ECG data from 100 healthy term babies for the first 24 hours after birth, to describe the trajectory of normal heartbeat variability in healthy term babies.

DATA ANALYSIS AND OUTCOME MEASURES

The prognostic accuracy (sensitivity, specificity, 95% confidence intervals) of early heartbeat variability using optimal cut-off values will be reported for the primary outcome. Logistic regression models adjusted for potential confounders will be used to report secondary outcomes.

POTENTIAL BENEFIT TO PATIENTS

Once the most accurate HRV indices and thresholds are identified, this data can be readily incorporated into a bed side real-time monitoring device. This device may have several clinical implications, including (i) improving access to treatment and the number of babies who benefit from being offered cooling; (ii) avoiding cooling therapy to low risk infants with hypoxic ischaemic encephalopathy (iii) maximising the therapeutic effect of cooling by reducing stress; (iv) enabling tailored neonatal nursing care based on real-time monitoring of neonatal stress and thus improving the long-term outcomes of babies with hypoxic ischaemic encephalopathy.

ELIGIBILITY:
HIE COHORT

Inclusion Criteria:

* Full term babies (>36 weeks)
* Requiring resuscitation at birth due to perinatal asphyxia and/or 5 minute Apgar score <6.
* Structured clinical neurological examination (modified Sarnat stage) within six hours of age suggestive of encephalopathy (mild, moderate or severe)
* Age less than six hours at the time of admission to the neonatal unit

Exclusion Criteria:

* Babies with lethal congenital malformations or cardiac conditions that could affect heartbeat variability
* Participation in any controlled trials of investigational medical products (C-TIMPS)

HEALTHY COHORT

Inclusion criteria:

* Healthy full term babies (>36 weeks) and birth weight between 9th to 91st centile
* Age less than six hours at the time of study enrolment

Exclusion criteria

* Babies requiring any medication or phototherapy
* Perinatal maternal fever

Ages: 0 Hours to 6 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Newborn babies within 6h of birth, healthy or with neonatal encephalopathy (mild, moderate or severe)
Sampling Method: Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2017-08-15 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2025-11-28 (Estimated)

PRIMARY OUTCOMES:
Prognostic accuracy of HRV to predict adverse neurodevelopment outcome | 18-22months
  Various linear and non-linear HRV indices will be compared with neurodevelopment at 18 to 22 months

SECONDARY OUTCOMES:
Correlation between HRV and salivary cortisol levels | first 5 days of live
  Various linear and non-linear HRV indices will be compared cortisol levels (measure of stress)

CONTACTS AND LOCATIONS:
Overall Officials: Sudhin Thayyil, Principal Investigator — Imperial College London
Locations (5):
- United Kingdom (5):
  - University Hospital Coventry & Warickshire NHS Trust, Coventry
  - Medway NHS Foundation Trust, Gillingham
  - Imperial College Healthcare NHS Trust, London
  - The Newcastle Upon Tyne NHS Foundation Trust, Newcastle
  - Norfolk & Norwich University Hospitals NHS Foundation Trust, Norwich

IPD SHARING:
Plan to Share IPD: No